CLINICAL TRIAL: NCT00058682
Title: A Phase III, Double Blind, Randomized, Multi-Center Study of the Safety and Efficacy of Anidulafungin VS. Fluconazole in the Treatment of Patients With Candidemia and Other Forms of Invasive Candidiasis and Prevention of Complications
Brief Title: Anidulafungin Versus Fluconazole in the Treatment of Candidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030150; 03-C-0150
Record Dates: First submitted 2003-04-11; First posted 2003-04-11 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-01

CONDITIONS: Candida; Candidiasis
Keywords: Fungal Infection; Mycoses; Candida Species; Candidiasis
MeSH Terms: conditions — Torulopsis; Candidiasis; Mycoses | interventions — Anidulafungin

INTERVENTIONS:
Drug: Anidulafungin

SUMMARY:
Fluconazole is an FDA-approved drug that is widely used to treat fungal infections due to candida. The experimental drug anidulafungin has been found to be active in treating life-threatening fungal infections. The purpose of this study is to determine whether anidulafungin is as effective as fluconazole in treating candidemia, an invasive form of candidiasis.

Three hundred patients 16 years of age or older will participate in this study. Participants will be randomly assigned to one of two groups: one-half will receive anidulafungin; the other half will receive fluconazole. They will receive the drug for as few as 10 days or for up to 42 days, depending on the seriousness of the infection. The drug will be given over a four-hour period on the first day, and over two hours on the remaining days. While taking the study medication, participants will be required to give blood samples every week until the end of treatment. At two weeks and six weeks following the end of therapy, participants will return for evaluation.

Prior to their participation in this study, patients will undergo the following evaluations: a physical exam, an eye exam, an electrocardiogram, and possibly blood work.

DETAILED DESCRIPTION:
This study is designed as a prospective, randomized, double-blind, non-inferiority, multi-center trial of the safety and efficacy of anidulafungin versus fluconazole in patients with candidemia or other forms of invasive candidiasis. The objective of this study is to determine if anidulafungin is at least as effective as fluconazole in the treatment of patients with a diagnosis of candidemia and/or other forms of invasive candidiasis. The secondary objectives are to compare the safety of the two study drugs and determine the efficacy for the prevention of late Candida infections in patients treated with anidulafungin versus fluconazole. Assuming 25% of patients will be unevaluable at the end of intravenous therapy, 248 patients will be enrolled to obtain a total of 222 evaluable patients. Patients older than 16 years of age with candidemia or invasive candidiasis will be randomized to receive either anidulafungin or fluconazole. Patients randomized to anidulafungin will receive an IV loading dose on day one of 200mg followed by 100mg once daily. Patients randomized to fluconazole will receive an IV loading dose on day one of 800mg followed by an IV daily dose of 400mg. Patients will be maintained on IV therapy for a minimum of 10 days to a maximum of 42 days. After 10 days of therapy, patients on either study drug may be treated on an ambulatory basis with oral fluconazole therapy.

ELIGIBILITY:
INCLUSION CRITERIA

Diagnosis of candidemia or other forms of invasive candidiasis from a blood culture or a culture specimen from a normally sterile site, the sample preferably having been taken within 96 hours before study entry. The diagnosis will be based on the following:

1. Candidemia: at least one blood culture positive for yeast (in the absence of other demonstrated foci of infection).
2. Other Forms of Invasive Candidiasis:

   * Positive culture for yeast from a specimen from a normally sterile site with or without a positive blood culture;
   * Positive yeast culture from a newly-placed drain in a normally sterile site; or
   * Any positive blood culture for yeast plus ophthalmic examination consistent with Candida endophthalmitis (patients with mycological documentation of Candida endophthalmitis with negative blood cultures will be included).
   * Positive yeast cultures from urine or sputum do NOT qualify as a positive culture.
3. AND at least one of the following signs and symptoms:

   * A fever defined as an oral temperature of 100.4° (Degree) F (38.0° (Degree)C) or greater, rectal temperature of 101.4° (Degree) F (38.4° (Degree)C) or greater, or an axillary temperature of 99.4° (Degree) F (37° (Degree)C) or greater. Hypothermia defined as a temperature less than 96.8° (Degree) F (36.0° (Degree)C).
   * A systolic blood pressure of less than 100 mmHg or a decrease in systolic blood pressure of at least 30 mmHg from patient's normal systolic blood pressure.
   * Some sign of inflammation (swelling, heat, erythema, purulence, or drainage from a wound) at a site positive for Candida
   * Signs or symptoms of candidemia/invasive candidiasis.
4. Radiological findings of invasive candidiasis.
5. Male or female 16 years of age or older.
6. Willing and able to give signed informed consent, or have a legally authorized representative who is willing and able to give consent. Informed assent will be required for children less than 18 years of age.
7. Reliable and willing to make themselves available for the duration of the study and to abide by the study restrictions.
8. Expected hospitalization of at least 3 days.

EXCLUSION CRITERIA

1. Female patients who are pregnant, lactating (breast feeding) or planning a pregnancy during the course of the study, or who are of child bearing potential and not using an acceptable method of birth control (i.e. abstinence, surgically sterile, intrauterine device, oral contraceptive plus barrier contraceptive, hormone delivery system plus barrier contraceptive or condom in combination with contraceptive cream, jelly or foam). Patients are to continue contraceptive methods during the study and for at least 30 days after receiving their last treatment.
2. Patients who have received greater than 72 hours of systemic antifungal therapy for the Candida infection for which they will be enrolled (patients who develop their Candida infection while receiving caspofungin or azole therapy will also be excluded).
3. Patients who have received prophylactic administration of fluconazole, itraconzaole, or voriconazole greater than or equal to one week within 30 days prior to enrollment.
4. Patients who have failed antifungal therapy with any systemic antifungal for this episode of candidiasis/candidemia. Recurrence within 2 weeks is considered failure of previous therapy.
5. Patients with suspected Candida osteomyelitis, endocarditis, or meningitis.
6. Patients with prosthetic devices which are a suspected site of infection are excluded unless the device is removed at study entry or soon after randomization. [Hemodialysis shunts (AV fistulae) may reamin in situ].
7. Patients with prosthetic heart valves or vascular grafts suspected to be the site of the candida infection and positive blood cultures.
8. Patients receiving and who will continue to receive terfenadine, cisapride, dofetilide, quinidine, pimozide and rifampin.
9. Patients who have, at any time, previously received anidulafungin.
10. Known Candida krusei infection.
11. Patients requiring continued treatment with another systemic antifungal agent [oral non-absorbable azoles (e.g., clotrimazole troches) are permitted].
12. Patients with a known hypersensitivity to echinocandin therapy or azole therapy.
13. Patients with any of the following abnormal laboratory values:

    1. bilirubin greater than 5 times theULN
    2. AST or ALT greater than 5 times theULN
14. Patients with poor venous access that would preclude intravenous drug delivery or multiple blood draws.
15. Patients who have participated in a study of an investigational drug or device (without any FDA approved indications) within four weeks of study entry. The investigational use of antiretroviral agents and the investigational use of licensed agents is permitted if the patient is on a stable regimen for four weeks prior to study start.
16. Life expectancy less than 72 hours.
17. Patients on hemodialysis unable to tolerate the volume of IV fluid on non-dialysis days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248
Dates: Start 2003-04; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wey SB, Mori M, Pfaller MA, Woolson RF, Wenzel RP. Hospital-acquired candidemia. The attributable mortality and excess length of stay. Arch Intern Med. 1988 Dec;148(12):2642-5. doi: 10.1001/archinte.148.12.2642. PMID 3196127
- [Background] Jarvis WR. Epidemiology of nosocomial fungal infections, with emphasis on Candida species. Clin Infect Dis. 1995 Jun;20(6):1526-30. doi: 10.1093/clinids/20.6.1526. PMID 7548503
- [Background] Pfaller MA. Epidemiology and control of fungal infections. Clin Infect Dis. 1994 Aug;19 Suppl 1:S8-13. doi: 10.1093/clinids/19.supplement_1.s8. PMID 7948573
- [Derived] Kett DH, Shorr AF, Reboli AC, Reisman AL, Biswas P, Schlamm HT. Anidulafungin compared with fluconazole in severely ill patients with candidemia and other forms of invasive candidiasis: support for the 2009 IDSA treatment guidelines for candidiasis. Crit Care. 2011;15(5):R253. doi: 10.1186/cc10514. Epub 2011 Oct 25. PMID 22026929
- [Derived] Reboli AC, Shorr AF, Rotstein C, Pappas PG, Kett DH, Schlamm HT, Reisman AL, Biswas P, Walsh TJ. Anidulafungin compared with fluconazole for treatment of candidemia and other forms of invasive candidiasis caused by Candida albicans: a multivariate analysis of factors associated with improved outcome. BMC Infect Dis. 2011 Sep 30;11:261. doi: 10.1186/1471-2334-11-261. PMID 21961941